CLINICAL TRIAL: NCT04962750
Title: Low Level Laser Therapy for Treatment of Tinnitus in Red Sea Scuba Divers: A Randomized Clinical Study
Brief Title: Low Level Laser Therapy for Treatment of Tinnitus in Red Sea Scuba Divers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N13476
Record Dates: First submitted 2021-07-03; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser therapy (Experimental)
  Interventions: Device: Low level laser therapy
- Control (Sham Comparator)
  Interventions: Other: Sham device

INTERVENTIONS:
Device: Low level laser therapy — Low level laser therapy from suitable machine
  Arms: laser therapy
Other: Sham device — The device wasn't working
  Arms: Control

SUMMARY:
Scuba Diving has become a popular hobby, for a leisure activity, diving puts the auditory system at the risk of a wide variety of complaints including tinnitus, Low level laser therapy is a new modality in treatment of tinnitus. This study evaluates effect of laser therapy on tinnitus of Scuba divers in Red Sea.

ELIGIBILITY:
Inclusion Criteria:

- scuba divers

Exclusion Criteria:

* Other ear or neurological diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Tinnitus Questionnaire score | 20 days
  A score that evaluates level of tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Osama El-sayyad, Principal Investigator — Benha University

IPD SHARING:
Plan to Share IPD: No